CLINICAL TRIAL: NCT01490502
Title: A Randomized Controlled Trial of Vitamin D Supplementation in Multiple Sclerosis
Brief Title: Vitamin D Supplementation in Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Oregon Health and Science University (Other); University of California, San Francisco (Other); Washington University School of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other); University of Pennsylvania (Other); Yale University (Other); The Cleveland Clinic (Other); University of Rochester (Other); Stanford University (Other); University of Virginia (Other); Swedish Medical Center (Other); Anne Arundel Health System Research Institute (Other); Columbia University (Other); University of Massachusetts, Worcester (Other); Dignity Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00049137
Record Dates: First submitted 2011-12-06; First posted 2011-12-13 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-dose vitamin D3 (Active Comparator)
  Interventions: Drug: Vitamin D3
- High-dose vitamin D3 (Active Comparator)
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Patients will be assigned to low dose (600 IU/day) versus high-dose (5000 IU/day) of vitamin D3 as an add-on therapy to glatiramer acetate (Copaxone).

SUMMARY:
Low vitamin D levels have been shown to increase a person's risk of developing multiple sclerosis (MS), and patients with MS who have lower vitamin D levels are at increased risk of having attacks. However, it is not known if giving supplemental vitamin D to those with MS reduces the risk of attacks, and some research suggests that vitamin D could even be harmful to people with MS.

In this clinical trial, patients with relapsing-remitting MS will receive high-dose or low-dose oral vitamin D in addition to an approved therapy for MS, glatiramer acetate. Patients will be evaluated for two years, and the effect of high-dose vitamin D supplementation on the rate of MS attacks and on the number of new lesions and change in brain volume on MRI will be determined. Establishing this association will have major implications for the treatment of individuals with MS throughout the world.

DETAILED DESCRIPTION:
Vitamin D insufficiency has recently emerged as a risk factor for susceptibility to multiple sclerosis (MS). The investigator's observational data suggest that lower vitamin D levels in patients with relapsing-remitting MS are associated with a higher subsequent relapse rate. However, it is unknown if providing vitamin D supplementation to such patients leads to a reduction in the risk of an exacerbation. Historically, several nutritional supplements that appeared to be helpful in observational studies of various diseases did not demonstrate a benefit or were harmful in randomized trials. Further, a vitamin D response element was recently identified in the promoter region of Human Leukocyte Antigen (HLA)-DRB1*15, the gene believed to be critical to initiating the autoimmune response in MS, and 1, 25-dihydroxyvitamin D3 increases the expression of the gene in vitro, suggesting that vitamin D supplementation could even be harmful in established MS.

This is a randomized, double-blind trial of high- versus low-dose vitamin D3 supplementation as an add-on to glatiramer acetate in 172 patients with relapsing-remitting MS. Subjects will be randomized to 600 IU or 5000 IU of oral vitamin D3 daily for two years. A standardized brain MRI scan will be performed at baseline and at the end of the first and second years. The impact of high-dose vitamin D supplementation on the number of relapses, the number of new lesions on brain MRI, and the change in brain volume will be assessed. Establishing these associations will have major implications for the treatment of patients with MS throughout the world and will provide rationale for further investigations of the role of vitamin D in the immunopathogenesis of MS, possibly leading to the identification of new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Must meet Magnetic Resonance Imaging in MS (MAGNIMS) criteria for relapsing-remitting MS
* Age 18 to 50 years
* Expanded Disability Status Scale (EDSS) score ≤ 4.0
* MS disease duration ≤ 10 years if McDonald Relapse Remitting Multiple Sclerosis (RRMS;) ≤ 1 year if meets MAGNIMS RRMS criteria but not McDonald RRMS criteria
* If the patient meets the McDonald RRMS criteria (rather than McDonald Clinically

Isolated Syndrome (CIS) that is now classified as MAGNIMS MS):

* Must have had one clinical attack in past two years and at least one new silent T2 or gadolinium-enhancing lesion on brain MRI within the past year OR
* Must have had two clinical attacks in past two years, one of which occurred in the past year
* Females of child-bearing age must be willing to use at least one form of pregnancy prevention throughout the study.
* Must have had a 25-hydroxyvitamin D level of ≥ 15 ng/mL within past 30 days
* Must be willing to stop taking additional supplemental vitamin D, except as part of a multivitamin, and must be willing to not take cod liver oil.

Exclusion Criteria:

* Not be pregnant or nursing
* No ongoing renal or liver disease
* No known history of nephrolithiasis, hypercalcemia, sarcoidosis or other serious chronic illness including cancer (other than basal cell or squamous cell carcinoma of the skin), cardiac disease, or HIV.
* No ongoing hyperthyroidism or active infection with Mycobacterium species
* No known gastrointestinal disease (ulcerative colitis, Crohn's disease, celiac disease/gluten intolerance) or use of medications associated with malabsorption.
* No history of self-reported alcohol or substance abuse in past six months.
* No prior history of treatment with rituximab, any chemotherapeutic agent, or total lymphoid irradiation. No treatment in the past six months with natalizumab, fingolimod, or fumarate. If patient has received glatiramer acetate, they have not been exposed to more than three months of treatment. No treatment with other unapproved therapies for MS.
* No use of interferon beta or glatiramer acetate therapy for one month prior to screening
* No use of more than 1,000 IU vitamin D3 daily in the three months prior to screening
* No condition that would limit the likelihood of completing the MRI procedures
* No use of thiazide diuretics, digoxin, diltiazem, verapamil, cimetidine, heparin, low-molecular weight heparin, phenytoin, phenobarbital, carbamazepine, routine corticosteroids (eg scheduled monthly steroids, daily, etc), rifampin, or cholestyramine.
* No steroids within a month of screening.
* Not suicidal at screening visit (ineligible if answers "yes" to question 1 of screening Columbia Suicide Severity Rating Scale (C-SSRS) in PAST 2 MONTHS; or answers "yes" to questions 2-5 on C-SSRS for PAST 6 MONTHS; or answers "yes" to suicidal attempts or preparatory attempts in PAST 5 YEARS , http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM225130.pdf).
* Serum calcium >0.2 mg/dL above upper limit of normal.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Mowry, MD, MCR, Principal Investigator — Johns Hopkins University
Locations (16):
- United States (16):
  - Dignity Health Medical Foundation, Carmichael, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Yale University, New Haven, Connecticut
  - Anne Arundel Health System Research Institute, Annapolis, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - Columbia University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Cassard SD, Fitzgerald KC, Qian P, Emrich SA, Azevedo CJ, Goodman AD, Sugar EA, Pelletier D, Waubant E, Mowry EM. High-dose vitamin D3 supplementation in relapsing-remitting multiple sclerosis: a randomised clinical trial. EClinicalMedicine. 2023 Apr 13;59:101957. doi: 10.1016/j.eclinm.2023.101957. eCollection 2023 May. PMID 37125397
- [Derived] Bhargava P, Cassard S, Steele SU, Azevedo C, Pelletier D, Sugar EA, Waubant E, Mowry EM. The vitamin D to ameliorate multiple sclerosis (VIDAMS) trial: study design for a multicenter, randomized, double-blind controlled trial of vitamin D in multiple sclerosis. Contemp Clin Trials. 2014 Nov;39(2):288-93. doi: 10.1016/j.cct.2014.10.004. Epub 2014 Oct 12. PMID 25311447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from March 2012 through April 2019 at 16 neurology clinics in the United States.
Pre-assignment Details: After successful screening, a thirty day run-in period was used to assess compliance with daily subcutaneous glatiramer acetate injections. Participants who missed more than 3 injections during the run-in period were ineligible to be randomized and were withdrawn from further study participation.
Period: Overall Study
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Started | 83 | 89
Received Allocated Intervention | 83 | 88
Attended at Least 1 Follow-up Visit | 82 | 83
Completed | 68 | 72
Not Completed | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3 | Total
Number analyzed (Participants) | 83 | 89 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (7.7) | 34.5 (7.1) | 34.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 61 | 131
  Male | 13 | 28 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 30
  Not Hispanic or Latino | 70 | 71 | 141
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 11 | 29
  White | 61 | 71 | 132
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 83 | 89 | 172
Expanded Disability Status Scale (EDSS) score [Median (Inter-Quartile Range); unit: units on a scale] — The Expanded Disability Status Scale (EDSS) is an ordinal clinical rating scale based on a standard neurological examination and is used to measure global neurologic impairment in people with multiple sclerosis (MS). It ranges from a minimum of 0.0 (normal examination) to 10.0 (death due to MS) in half-point increments. Population: Screening EDSS was used for one high-dose vitamin D3 participant with missing EDSS at baseline.
  units on a scale | 2.00 [1.00 to 2.50] | 2.00 [1.50 to 2.50] | 2.00 [1.38 to 2.50]
Multiple Sclerosis Functional Composite (MSFC) score [Mean (Standard Deviation); unit: Z-score] — The Multiple Sclerosis Functional Composite (MSFC) is a three-part measure of disability for people with multiple sclerosis, including measures of leg function/ambulation, arm/hand function and cognitive function. The three independent measures have different units. We take the reciprocal of the arm/hand function test, and then convert all measures to Z-scores. The average of the Z-scores from each measure yields the MSFC composite Z-score. A Z-score of 0 represents the population mean and positive scores indicate less disability.
  Z-score | 0.5 (0.4) | 0.6 (0.5) | 0.5 (0.4)
Low-contrast acuity [Mean (Standard Deviation); unit: letters] — Low-contrast acuity was measured as binocular vision on a 2.5% Sloan chart at a distance of 2 meters. The chart is used to test the ability to discriminate gradually smaller gray letters with a 2.5% contrast level against a white background. The low-contrast acuity measure is scored as total letters read and ranges from 0 (no letters read) to 60 (all letters read), with higher scores indicating better low-contrast acuity.
  letters | 36 (10) | 34 (10) | 35 (10)
Health-related Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The Functional Assessment of Multiple Sclerosis (FAMS) is the quality of life (QOL) instrument used in this trial. It consists of 44 questions and the total score has a possible range of 0 to 176, with higher scores indicating better QOL.
  units on a scale | 126 (24) | 126 (27) | 126 (26)
Normalized Brain Parenchymal Volume [Mean (Standard Deviation); unit: microliters] — Population: Baseline Brain MRI not available or not of sufficient quality to compute measure for 9 low-dose vitamin D3 and 7 high-dose vitamin D3 participants.
  microliters
    number analyzed (Participants) | 74 | 82 | 156
    (all) | 1,488,270 (107,046) | 1,496,147 (88,025) | 1,492,411 (97,270)
Normalized Gray Matter Volume [Median (Inter-Quartile Range); unit: microliters] — Population: Baseline Brain MRI not available or not of sufficient quality to compute measure for 9 low-dose vitamin D3 and 7 high-dose vitamin D3 participants.
  microliters
    number analyzed (Participants) | 74 | 82 | 156
    (all) | 772,736 [735,433 to 809,191] | 781,461 [737,843 to 807,965] | 774,469 [736,684 to 808,542]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects That Experience a Relapse
Description: Confirmed relapse defined as new or worsening symptoms referable to the central nervous system, lasting at least 24 hours, occurring at least 30 days since the prior attack, accompanied by worsening of the EDSS (>= 0.5 points) or in the Functional Systems (FS) scales (2 points on at least one FS scale or 1 point on >= two FS scales).
Time Frame: 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
proportion of participants | 0.32 | 0.34
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.60, Log Rank
Statistical Analysis 2: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.57, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.67 to 2.05]

2. Secondary Outcome: Annualized Relapse Rate
Description: Average relapses per year
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: relapses per participant per year
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
relapses per participant per year | 0.20 [0.11 to 0.35] | 0.34 [0.20 to 0.56]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Other; p = 0.07, Andersen Gill model for recurrent events

3. Secondary Outcome: Number of Relapses Requiring Treatment
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: relapses
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
relapses | 0.15 [0.08 to 0.30] | 0.28 [0.15 to 0.51]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.07, Negative Binomial Model; Rate Ratio = 1.80, 95% CI 2-sided [0.94 to 3.45]

4. Secondary Outcome: Number of New or Enlarging T2 Lesions
Time Frame: 2 years
Population: Participants analyzed had > 1 MRI during the study (baseline and at least one follow-up MRI of sufficient quality).
Measure: Mean (95% Confidence Interval); unit: lesions
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 65 | 74
lesions | 1.95 [1.16 to 3.29] | 2.88 [1.78 to 4.64]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.14, Negative Binomial Model; Rate Ratio = 1.47, 95% CI 2-sided [0.88 to 2.46]

5. Secondary Outcome: Proportion of Participants With Sustained Disability Progression
Description: The Expanded Disability Status Scale (EDSS) is an ordinal clinical rating scale based on a standard neurological examination and is used to measure global neurologic impairment in people with multiple sclerosis (MS). It ranges from a minimum of 0.0 (normal examination) to 10.0 (death due to MS) in half-point increments. A participant will be considered to have had sustained progression of disability if there is an increase in the EDSS score at month 12 by at least 1.0 point that is confirmed on the final examination one year later (month 24).
Time Frame: 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
proportion of participants | 0.05 | 0.08
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.60, Log Rank

6. Secondary Outcome: Change in Multiple Sclerosis Functional Composite (MSFC) Score
Description: The Multiple Sclerosis Functional Composite (MSFC) is a three-part measure of disability for people with multiple sclerosis, including measures of leg function/ambulation, arm/hand function and cognitive function. The three independent measures have different units. We take the reciprocal of the arm/hand function test, and then convert all measures to Z-scores. The average of the Z-scores from each measure yields the MSFC composite Z-score. A Z-score of 0 represents the population mean and positive scores indicate less disability.
  The MSFC was measured at baseline and up to 4 more times over 2 years.
Time Frame: 2 years
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
Z-score | 0.051 [0.022 to 0.079] | 0.025 [-0.003 to 0.053]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; The average rate of change in MSFC Z-score over time was analyzed using a linear mixed-effects model with unstructured covariance structure and random intercepts. The p-value is a test of whether there is a difference in the rate of change in the MSFC Z-score between treatment arms; Test type: Superiority; p = 0.20, Mixed Models Analysis

7. Secondary Outcome: Change in Low-contrast Acuity
Description: Low-contrast acuity was measured as binocular vision on a 2.5% Sloan chart at a distance of 2 meters. The chart is used to test the ability to discriminate gradually smaller gray letters with a 2.5% contrast level against a white background. The low-contrast acuity measure is scored as total letters read and ranges from 0 (no letters read) to 60 (all letters read). Low-contrast acuity was measured at baseline and up to 4 more times over 2 years and higher scores indicate better low-contrast acuity.
Time Frame: 2 years
Population: Participants analyzed did not have an MS relapse between screening and baseline visits and had at least one low-contrast acuity measure at a follow-up visit.
Measure: Mean (95% Confidence Interval); unit: letters
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 79 | 78
letters | 0.82 [-0.08 to 1.71] | 1.09 [0.20 to 1.99]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Rate of change in 2.5% low-contrast acuity was analyzed using a linear mixed effects model with unstructured covariance structure and random intercepts. The p-value is a test of whether there is a difference in the rate of change in low-contrast acuity between treatment arms; Test type: Superiority; p = 0.67, Mixed Models Analysis

8. Secondary Outcome: Change in Health-related Quality of Life
Description: The Functional Assessment of Multiple Sclerosis (FAMS) questionnaire is the quality of life (QOL) instrument used in this trial. It consists of 44 questions and the total score has a possible range of 0 to 176, with higher scores indicating better QOL. The FAMS questionnaire was obtained at baseline and up to 4 more times over 2 years.
Time Frame: 2 years
Population: Participants analyzed completed a baseline FAMS questionnaire and at least 1 follow-up FAMS questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 79 | 78
score on a scale | -0.78 [-2.38 to 0.82] | -2.21 [-3.81 to -0.62]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Rate of change in quality of life was analyzed using a linear mixed effects model with unstructured covariance structure and random intercepts. The p-value is a test of whether there is a difference in the rate of change in health-related quality of life between treatment arms; Test type: Superiority; p = 0.21, Mixed Models Analysis

9. Secondary Outcome: Change in Brain Parenchymal Volume
Time Frame: 2 years
Population: Participants analyzed had > 1 MRI during the study (baseline MRI and at least one follow-up MRI of sufficient quality).
Measure: Mean (95% Confidence Interval); unit: microliters
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 65 | 74
microliters | -0.29 [-0.78 to 0.20] | -0.81 [-1.28 to -0.34]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.13, Mixed Models Analysis

10. Secondary Outcome: Change in Normalized Gray Matter Volume
Time Frame: 2 years
Population: Participants analyzed had > 1 MRI during the study (baseline MRI and at least one follow-up MRI of sufficient quality).
Measure: Mean (95% Confidence Interval); unit: microliters
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 65 | 74
microliters | -0.15 [-0.73 to 0.45] | -0.87 [-1.43 to -0.31]
Statistical Analysis 1: Comparison: Low-dose Vitamin D3 vs High-dose Vitamin D3; Test type: Superiority; p = 0.08, Mixed Models Analysis

11. Secondary Outcome: Change in Cortical Thickness
Description: Unable to analyze this outcome measure
Time Frame: 2 years
Population: The quality of the clinical MRI scans acquired for this study prevented the analysis of cortical thickness.
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Development of Hypercalcemia
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
Participants | 0 | 0

13. Secondary Outcome: Development of Nephrolithiasis
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
Number analyzed (Participants) | 82 | 83
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Low-dose Vitamin D3 | High-dose Vitamin D3
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 11/82 | 11/83
Other Adverse Events (participants affected / at risk) | 66/82 | 63/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Vitamin D3 (N=82) | High-dose Vitamin D3 (N=83)
Hypercalcemia (Endocrine disorders) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Unplanned pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 (6) | 3 (3)
Unplanned hospitalization (Nervous system disorders) | 1 (1) | 3 (7)
Unplanned hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5)
Unplanned hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Unplanned hospitalization (Psychiatric disorders) | 1 (2) | 0 (0)
Unplanned hospitalization (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Unplanned hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unplanned hospitalization (Eye disorders) | 0 (0) | 1 (1)
Planned hospitalization for elective procedure (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Planned hospitalization for elective procedure (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Planned hospitalization for elective procedure (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Vitamin D3 (N=82) | High-dose Vitamin D3 (N=83)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 28 (44) | 26 (40)
Numbness or tingling (Nervous system disorders) | 20 (22) | 20 (21)
Headache / worsened headache / migraine (Nervous system disorders) | 13 (14) | 18 (22)
Fatigue / increased fatigue (Nervous system disorders) | 14 (14) | 11 (11)
Joint pain or swelling (Musculoskeletal and connective tissue disorders) | 7 (10) | 11 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 7 (7)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 4 (5)
Depression / increased depression / severe depression (Psychiatric disorders) | 6 (6) | 9 (10)
Influenza (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Abdominal pain / cramp / discomfort (Gastrointestinal disorders) | 8 (8) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4)
Limb pain (Nervous system disorders) | 4 (6) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Urinary tract infection (Renal and urinary disorders) | 7 (7) | 2 (3)
Urinary dysfunction (Renal and urinary disorders) | 3 (3) | 4 (6)
Dizziness / increased dizziness (Ear and labyrinth disorders) | 4 (4) | 5 (5)
Spasm / cramp (non-abdominal) (Nervous system disorders) | 3 (3) | 6 (6)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Anxiety / worsening anxiety (Psychiatric disorders) | 3 (3) | 5 (6)
Sleep disorder (Psychiatric disorders) | 5 (5) | 11 (11)
Sore throat (+/- streptococcal infection) (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT01490502/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT01490502/SAP_001.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT01490502/ICF_002.pdf